CLINICAL TRIAL: NCT02821325
Title: Intra-articular Volumetric Assessment After Total Knee Arthroplasty
Acronym: TKA
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Principal Investigator, Nirav Amin, MD, Associate Professor, Loma Linda University
Other Study IDs: 5160043
Record Dates: First submitted 2016-04-25; First posted 2016-07-01 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Hematoma
MeSH Terms: conditions — Hematoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MRI: Radiology
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Patients undergoing a total knee arthroplasty, will undergo additional MRI's. One MRI pre-operatively.
  2nd MRI post-operatively on day 1. 3rd MRI post-operatively on day 2.

SUMMARY:
The purpose of the study: is to quantify the amount of post-operative effusion or hematoma present after total knee arthroplasty pre-operatively, post-operative day #0,1.

Patients undergoing a total knee arthroplasty will undergo an MRI on the operative knee at the following times:

* Pre-operatively
* Post-operative day #1 (approximately 16-20 hours post op)
* Post-operative day #2 (approximately 36-40 hours post op) This will be conducted by the Loma Linda radiology department as per normal protocols. No special imaging procedures will be undertaken.

Subjects will be both male and females, they will be patients from the Principle Investigator and Co-Investigators practice. Subjects will be between the ages of 18-89 years of age.

The total participation will last approximately 30 days.

Subject selection will be approximately 10 English speaking, both male and female between the ages of 18 to 89 years of age. Subjects will be recruited from the Principal Investigators and Co-Investigators clinic. There will be no advertising or electronic recruiting. The study is expected to last 12 months.

DETAILED DESCRIPTION:
STUDY DESIGN:

Background or rationale for this study:

Total knee arthroplasty is one of the most successful orthopedic surgeries performed in the United States, and consistently has shown to have excellent outcomes for patients, with low complication rates. However, when complications do happen, they can range from superficial infection to repeated deep infection requiring prosthesis exchange or amputation. Another significant complication of total knee arthroplasty is joint stiffness. Range of motion loss can also be an extremely debilitating complication necessitating prolonged physical therapy, return to the operating theater for manipulation or even total synovectomy and polyethylene exchange.

Although it is currently known that post-operative hematoma leads to adverse outcomes following total knee arthroplasty, there is currently no literature to quantify the average size or progression of the intra-articular bleeding post operatively. It would be reasonable to assume that all patients develop a slight hematoma post operatively. The investigator aims to assess the size, and possible progression of the intra-articular hematoma following total knee arthroplasty.

OBJECTIVES:

The investigator aims to:

Quantify the amount of post-operative effusion or hematoma present after total knee arthroplasty pre-operatively, post-operative day #0, 1.

Procedures involved (Research Interventions)

Patients undergoing a total knee arthroplasty will undergo an MRI of the operative knee at the following times:

* Pre-operatively
* Post-operative day #1 (approximately 16-20 hours post op)
* Post-operative day #2 (approximately 36-40 hours post op)

This will be conducted by the Loma Linda radiology department as per normal protocols. No special imaging procedures will be undertaken.

No changes in operative technique or post-operative protocol will be undertaken due to study apart from the above imaging.

All imaging will be kept on the LLUMC PACS system. Concise review of literature that supports the rationale, objectives, and methodology of the proposed study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective primary total knee arthroplasty.
* Patients not meeting exclusion criteria

Exclusion Criteria:

* If patient is not able to undergo MRI
* Heart pacemaker
* Cochlear implant
* Metallic foreign body (metal silver) in the eyes
* Aneurysm clip in the brain
* Patient with prior reaction or contra-indication to tranexamic acid
* Inability to comprehend consent process
* Age <18 or > 89
* Patient planned for outpatient procedure
* Active malignancy
* Patients with hematologic disorders (hemophilia, factor V Leiden, etc.)
* Patients with any condition that makes undergoing a MRI painful (severe spine degenerative disease, vertigo, etc.)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that will undergoing a Total Knee Arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Participants with total knee arthroplasty assessed for intra-articular hematoma | 30 days
  MRI studies will be reviewed on these participants pre-operatively and postoperatively. Data will be analyzed using the Statistical package for social sciences (SPSS) software and paired T-Test will be utilized for significance regarding the effusion post operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Nirav H. Amin, MD, Principal Investigator — Loma Linda University Faculty
Locations (1):
- Loma Linda University Healthcare Department of Orthopaedic Surgery, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Sex and gender. The size of the implant placed during the TKA. Indication for operative procedure. Laterality of the procedure. Operative time. Blood Loss from surgery. Range of motion at week 2 post-operatively. Range of motion at week 6 post-operatively. Any complications that develop within 30 days of the surgery. There is no plan to make individual participant data available.